CLINICAL TRIAL: NCT00276887
Title: Cognitive Behavior Therapy for Somatization Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K08MH001662 (NIH); K08MH001662 (NIH); DSIR AT-CD
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Somatoform Disorders
Keywords: Somatization Disorder; Multiple Medically Unexplained Symptoms; Cognitive Behavior Therapy; Mental Health
MeSH Terms: conditions — Somatoform Disorders; Psychological Well-Being | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy
Behavioral: Psychiatric Consultation Letter

SUMMARY:
This study will examine the long-term effects of cognitive behavioral therapy on the physical symptoms, functioning, and health care utilization of people with multiple medically unexplained physical symptoms.

DETAILED DESCRIPTION:
Somatization disorder is a chronic psychological condition that causes numerous physical complaints for which no underlying physical problem can be identified. The disorder often lasts for several years and results in substantial functional impairment. The physical complaints most frequently involve chronic pain and problems with the digestive, nervous, and reproductive systems. Neither pharmacological nor psychosocial treatments for this disorder have been successful in suppressing symptoms. Cognitive behavioral therapy (CBT) is a treatment that focuses on maladaptive patterns of thinking and the beliefs that underlie such thinking. This study will examine the long-term effects of CBT on the physical symptoms, functioning, and health care utilization of people with somatization disorder.

Participants in this open label study will be randomly assigned to receive either CBT supplemented with augmented standard medical care (ASMC) as indicated by a psychiatric consultation letter or ASMC alone. Participants assigned to CBT plus ASMC will receive CBT for 10 weeks. Somatic symptomatology, functional impairment, and health care costs will be assessed at study visits at baseline and Months 3, 9, and 15. The visits at Months 9 and 15 will assess specifically the long-term efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for somatization disorder
* Available for follow-up over the ensuing 15 months
* English-speaking

Exclusion Criteria:

* Meets DSM-IV criteria for a psychotic disorder, organic brain syndrome, or psychoactive substance dependence
* Active suicidal ideation
* Unstable major medical condition
* Plans to engage in additional psychotherapy during the first 3 months after study entry
* Current use of any medication that has not been stabilized for the 2 months prior to study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 1999-09; Primary Completion 2003-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Symptoms of somatization disorder
Functioning (measured with the Clinical Global Impression Scale for Somatization Disorder at Months 9 and 15)

SECONDARY OUTCOMES:
Health care utilization (measured the year before baseline and during the year after the 3-month assessment)
Health status (measured by the Medical Outcomes Study, SF-36, at Months 9 and 15)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley A. Allen, PhD, Principal Investigator — University of Medicine & Dentistry of New Jersey - Robert Wood Johnson Medical School
Locations (1):
- Department of Psychiatry, UMDNJ - RWJ Medical School, Piscataway, New Jersey, United States

REFERENCES:
- [Background] Allen LA, Woolfolk RL, Lehrer PM, Gara MA, Escobar JI. Cognitive behavior therapy for somatization disorder: a preliminary investigation. J Behav Ther Exp Psychiatry. 2001 Jun;32(2):53-62. doi: 10.1016/s0005-7916(01)00020-9. PMID 11764061
- [Background] Allen LA, Escobar JI, Lehrer PM, Gara MA, Woolfolk RL. Psychosocial treatments for multiple unexplained physical symptoms: a review of the literature. Psychosom Med. 2002 Nov-Dec;64(6):939-50. doi: 10.1097/01.psy.0000024231.11538.8f. PMID 12461199